CLINICAL TRIAL: NCT00844688
Title: A Phase II Feasibility Study of Sorafenib and Gemcitabine Combination Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Sorafenib and Gemcitabine in Advanced Hepatocellular Carcinoma (HCC)
Acronym: HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Collaborators: Bayer (Industry)
Responsible Party: Colonel Naeem Naqi, Combined Military Hospital, Rawalpindi, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; Gemcitabine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib/gemcitabine (Other)
  Interventions: Drug: sorafenib; Drug: Gemcitabine

INTERVENTIONS:
Drug: sorafenib — Patients will be treated with 400 mg oral sorafenib twice a day on a continuous basis. Patients in this protocol may continue to be treated with this combination for a minimum of 4 cycles until any of the following criteria for protocol discontinuation is reached:
  1. Progression of disease.
  2. The patient is unlikely to benefit from further treatment as
     Judged by the Investigator.
  3. Intolerable toxicity of the drugs.
  4. Withdrawal of consent for any reason.
  Other Names: Nexavar
Drug: Gemcitabine — Patients will be treated with Gemcitabine 1000mg/m2 administered on day 1 & 8 of a 4 week cycle. Patients in this protocol may continue to be treated with this combination for a minimum of 4 cycles until any of the following criteria for protocol discontinuation is reached:
  Progression of disease. The patient is unlikely to benefit from further treatment as
  Judged by the Investigator.
  Intolerable toxicity of the drugs. Withdrawal of consent for any reason.
  Other Names: Gemzar

SUMMARY:
For the majority of patients, metastatic HCC is incurable and patients should be considered candidates for clinical trials when appropriate. Till recently there was no worldwide, approved local or systemic therapy for advanced HCC and the available therapies for advanced unresectable and/or metastatic HCC have limited clinical values, with low response rates and little impact on the natural history of the disease. Furthermore, the toxicities associated with these agents can be severe, requiring careful patient selection, and this dramatically decreases the number of patients who may benefit from therapy. The SHARP trial established the survival benefit of Sorafenib in Advanced HCC but the results yet remain humble. The need for more effective therapies is still there.

Study Objectives

The primary objective of this phase II study is to evaluate the efficacy and safety of Sorafenib and Gemcitabine combination in patients with advanced HCC.

Safety data and limited efficacy data will be collected for this combination in the study. All Drug-Related Adverse Events, all Adverse Events NCI CTCAE Version 3.0 Grade 3 or higher, and all Serious Adverse Events regardless of causal relationship to study drugs will be recorded in this study.

DETAILED DESCRIPTION:
Over-all Study Design

This is a non-randomized, open-label treatment protocol for patients with advanced HCC.

30 Patients will be treated with 400 mg oral sorafenib twice a day on a continuous basis with Gemcitabine 1000mg/m2 administered on day 1 & 8 of a 4 week cycle. Patients in this protocol may continue to be treated with this combination for a minimum of 4 cycles until any of the following criteria for protocol discontinuation is reached:

1. Progression of disease.
2. The patient is unlikely to benefit from further treatment as

   Judged by the Investigator.
3. Intolerable toxicity of the drugs.
4. Withdrawal of consent for any reason.

Dosage, administration and duration

Doses of study drugs may be delayed or reduced in case of clinically significant toxicities that are possibly, probably or definitely related to protocol therapy. Toxicities will be graded using the NCI Common Terminology Criteria Version 3.0 (see Appendix 10.6). If a patient experiences several toxicities and there are conflicting recommendations, the recommended dose adjustment that reduces the dose to the lowest level should be used. All dose modifications will follow pre-defined dose levels as indicated below for study drugs, respectively. The dose modifications of sorafenib will follow the following dose levels:

Dose level 1 (starting dose): 400 mg (2 x 200 mg) p. o. twice daily Dose level 2: 400 mg (2 x 200 mg) p. o. once daily Dose level 3: 400 mg (2 x 200 mg) p. o. once every other day If a dose reduction by more than two dose levels from the 400 mg twice daily schedule is required, the patient should be discontinued from the study treatment. Also, at the discretion of the Investigator, the dose may be re escalated to a higher dose level up to up to a maximum of 400 mg twice daily following the resolution of the Adverse Event or an improvement in the Adverse Event to a level which permits the re-escalation of the study drug.

For Gemcitabine the potentially dose limiting toxicity is myelosuppression, dose delays are allowed for Grade 3 and 4 toxicities. Growth factors will not be administered unless delay is more than 2 weeks in recovery of hematological toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced Hepatocellular carcinoma
2. Histologically proven
3. Child-Pugh A and B
4. Age > 18 years.
5. ECOG Performance Status of 0 or1
6. Life expectancy of at least 12 weeks.
7. Subjects with at least one uni-dimensional (for RECIST) or bi-dimensional (for WHO) measurable lesion. Lesions must be measured by CT-scan or MRI
8. Adequate bone marrow, liver and renal function as assessed by the following

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) >1,500/mm3
   * Platelet count ³ 100,000/μl
   * Total bilirubin < 1.5 times the upper limit of normal
   * ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
   * Alkaline phosphatase < 4 x ULN
   * PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
   * Serum creatinine < 1.5 x upper limit of normal. (normal creatinine value: 0.8-1.2 mg/dl)
   * Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or Digoxin are permitted) or uncontrolled hypertension.
2. History of HIV infection
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. History of organ allograft however, the organ allograft may be allowed as protocol specific.
7. Patients with evidence or history of bleeding diasthesis
8. Patients undergoing renal dialysis
9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.

Excluded therapies and medications, previous and concomitant:

1. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
2. Major surgery within 4 weeks of start of study
3. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
4. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
5. Prior exposure to the study drug.
6. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial (and men for at least 3 months after last administration of study medication). Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
7. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
RECIST criteria for response evaluation by CT sacan abdomen in Target lesion of HCC | 4 months

SECONDARY OUTCOMES:
Toxicity evaluation in accordance with CTCAE v3.0 | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Naqi, MBBS,FCPS, Principal Investigator — Consultant Oncologist
Locations (1):
- Combined Military Hospital, Rawalpindi, Punjab Province, Pakistan